CLINICAL TRIAL: NCT04737603
Title: Feasibility of Pediatric Emergency Department-Initiated Treatment for Adolescents With Opioid Use Disorder
Acronym: PEDsTREATOUD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was not funded and therefore not recruiting. So we never opened the study.
Sponsor: University of California, Davis (Other)
Collaborators: Yale University (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1707330
Record Dates: First submitted 2021-01-22; First posted 2021-02-04 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Opioid-use Disorder
Keywords: Buprenorphine; Adolescents; Pediatrics; Emergency Department
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies | interventions — Buprenorphine; Naloxone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ED-initiated treatment with buprenorphine/naloxone. (Experimental): A Clinical Opiate Withdrawal Score (COWS) score will be administered, and an induction dose of buprenorphine when COWS scores >=8. Participants who weigh > 70 kg and/or reported using ≥ 3 bags of heroin/day or its prescription opioid equivalent will receive 4 mg. After 1 hour an additional 4 mg will be administered for a total of 8 mg. Participants who weigh <= 70 kg and/or reported using ≤ 3 bags of heroin/day or its prescription opioid equivalent will receive 4 mg of buprenorphine. After 1 hour, an additional 2 mg will be administered for a total of 6 mg. Patients will be prescribed sufficient take-home daily doses (one-week supply) to ensure that the patient has adequate medication to receive 12-16 mg buprenorphine sublingual once daily. Parents of adolescents will also receive appropriate education on how to administer medication. Home induction instructions will be provided to patients and parents that arrive to the ED after an opioid overdose.
  Interventions: Drug: ED-Initiated treatment with buprenorphine / naloxone

INTERVENTIONS:
Drug: ED-Initiated treatment with buprenorphine / naloxone — A Clinical Opiate Withdrawal Score (COWS) score will be administered, and an induction dose of buprenorphine when COWS scores >=8. Participants who weigh > 70 kg and/or reported using ≥ 3 bags of heroin/day or its prescription opioid equivalent will receive 4 mg. After 1 hour an additional 4 mg will be administered for a total of 8 mg. Participants who weigh <= 70 kg and/or reported using ≤ 3 bags of heroin/day or its prescription opioid equivalent will receive 4 mg of buprenorphine. After 1 hour, an additional 2 mg will be administered for a total of 6 mg. Patients will be prescribed sufficient take-home daily doses (one-week supply) to ensure that the patient has adequate medication to receive 12-16 mg buprenorphine sublingual once daily. Parents of adolescents will also receive appropriate education on how to administer medication. Home induction instructions will be provided to patients and parents that arrive to the ED after an opioid overdose.
  Other Names: Suboxone

SUMMARY:
ED-initiated buprenorphine with brief intervention and facilitated referral to treatment has been shown to be highly successful in increasing treatment engagement rates and reducing opioid use among adults. It is unknown whether this intervention is similarly effective for adolescents with OUD. To rigorously examine this important clinical research question, it is first necessary to optimize this intervention for the adolescent population. In this R34 proposal, we will use the Assessment-Decision-Administration-Production-Topic Experts-Integration-Training-Testing (ADAPT-ITT) framework-a systematic method for intervention adaptation- to adapt (Aim 1) and test the feasibility (Aim 2) of a treatment strategy for adolescents that has been shown to effectively link adults with OUD to ongoing addiction treatment.

DETAILED DESCRIPTION:
The opioid epidemic is a serious public health crisis that affects all age groups. Emergency departments (EDs) are on the front line of this public health crisis. Buprenorphine is an Opioid Use Disorder (OUD) treatment that reduces opioid overdose mortality by up to 70%. A landmark 2015 randomized controlled trial (RCT) also demonstrated effectiveness of ED-initiated buprenorphine in improving OUD treatment engagement rates in adults. As a result, EDs across the nation have begun to follow these practices. This model of evidence-based treatment is a paradigm shift for care delivery and ripe for adaptation to special populations, such as adolescents. Adolescents with OUD need easy access to treatment now more than ever: fentanyl use is on the rise, the COVID-19 pandemic has heralded historic levels of social isolation in this age group, and the opioid overdose death rate is increasing.

Little research has examined how the ED can engage adolescents and their families in effective OUD treatment. Buprenorphine is an evidence-based treatment for OUD in adolescents. Three RCTs in ambulatory settings have demonstrated the efficacy of buprenorphine in reducing opioid use and improving treatment retention in adolescents with OUD. Given its efficacy, the American Academy of Pediatrics (AAP) recommends that pediatricians offer buprenorphine to adolescents with severe OUD or discuss referrals to other providers for this service. Despite the immense efforts to improve access to buprenorphine, youth with OUD continue to have markedly low rates of receiving this life-saving medication. A study of Medicaid-enrolled adolescents with OUD found that between 2014 and 2015, only 3.3% of 13-15 year-old and 6.9% of 16-17 year-old patients received OUD treatment medication within 3 months of diagnosis. Treatment receipt is even lower among adolescents experiencing opioid overdose; only 0.5% of 13-15 year-old and 0.8% of 16-17 year-old adolescents receive pharmacotherapy within 30 days of the overdose. Research is urgently needed to identify effective strategies to address the enormous treatment gap for adolescents with OUD.

ED-initiated buprenorphine with brief intervention and facilitated referral to treatment has been shown to be highly successful in increasing treatment engagement rates and reducing opioid use among adults. It is unknown whether this intervention is similarly effective for adolescents with OUD. To rigorously examine this important clinical research question, it is first necessary to optimize this intervention for the adolescent population. In this R34 proposal, we will use the Assessment-Decision-Administration-Production-Topic Experts-Integration-Training-Testing (ADAPT-ITT) framework-a systematic method for intervention adaptation- to adapt (Aim 1) and test the feasibility (Aim 2) of a treatment strategy for adolescents that has been shown to effectively link adults with OUD to ongoing addiction treatment. We aim to:

Aim 1: Optimize the intervention of ED-initiated buprenorphine with brief intervention and facilitated referral to treatment for adolescents (ages 13 years old until their 18th birthdays) with OUD (Year 1). Recognizing the novelty of ED-initiated treatment for OUD in adolescents, and the importance of ensuring that the evidence-based intervention components are relevant to the target population, we will use the ADAPT-ITT framework to systematically refine the intervention. Focus groups and in-depth interviews with key stakeholders will examine: 1) perceptions of ED-initiated buprenorphine, brief intervention and facilitated referral to treatment for adolescents, 2) preferences for content and delivery of the intervention, and 3) strategies to increase awareness and acceptability of the ED as an access site for treatment and linkage to care for adolescents. Data will be used to adapt intervention for EDs that treat adolescents and inform the development of updated intervention training protocols.

Aim 2. Conduct a single-arm pilot study of the intervention developed in Aim 1 to examine the feasibility of enrolling and collecting outcomes from adolescents (ages 13 years-old until their 18th birthdays) with OUD presenting to 4 pediatric EDs (Year 2). We will conduct this pilot study in 4 geographically diverse EDs within the Pediatric Emergency Care Applied Research Network (PECARN). PECARN is the only federally-funded pediatric emergency medicine research network with the robust infrastructure to identify and efficiently enroll a sufficient number of adolescents with OUD into an ED-based clinical trial. We hypothesize:

Hypothesis 1: We will enroll adolescents with OUD at a recruitment rate of at least 1 patient/site/month.

Hypothesis 2: We will retain 80% of participants at 30 days, as defined by the successful collection of the 30-day outcomes of treatment engagement, self-report of opioid use in the previous 7 days and urine toxicology for opioids.

Impact: The findings will inform our planned large-scale implementation trial of ED-initiated treatment in adolescents which could improve outcomes and ultimately save the lives of numerous U.S adolescents. The ADAPT-ITT process and feasibility study directly responds to an urgent need to design and test developmentally-appropriate OUD treatment engagement strategies for this age group.

ELIGIBILITY:
Inclusion Criteria:

1. 13 years-old up to their 18th birthday on day of enrollment
2. Meet DSM-5 criteria for moderate/severe opioid use disorder;
3. Have a urine toxicology test positive for opioids, oxycodone, or buprenorphine (non-prescribed by history)
4. Can provide information for 2 reliable contacts that the study staff can contact in the case the study participant cannot be reached

Exclusion Criteria:

1. Have a urine toxicology test positive for methadone;
2. Unable to provide consent due to critical illness or reduced capacity
3. In jail/prison or in police custody;
4. Under the guardianship of child protective services;
5. Requires opioid medications for a currently present chronic pain condition;
6. Transferred from the ED to an inpatient unit prior to being able to provide consent;
7. Already enrolled in formal OUD treatment with medications with intent to return to the treatment program after ED discharge; or
8. Previously enrolled in the current study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment engagement | 30 days
  Number of enrolled participants who 1) provide written consent for treatment status verification, 2) provide a urine toxicology sample. Reasons for not providing consent/toxicology sample will be recorded.
Mean number of days of self-reported opioid use as assessed by Timeline Follow-Back (TLFB) | 30 days
  Timeline Follow-Back (TLFB): The TLFB procedure will be used to elicit the patient participant's self- reported use, quantity, and route of administration of opioids, alcohol, tobacco, marijuana, stimulants, and benzodiazepines over the previous 7 days. The validity of adolescent self-report data on substance use and TLFB has been documented previously in the literature.
% of urine samples testing negative for opioid use | 30 days
  Patients will provide a urine sample at 30 days and will be tested for the presence of opioids.